CLINICAL TRIAL: NCT05579860
Title: A Single-Dose, Randomized, Open-Label, Two-Period Crossover, Bioequivalence Study Comparing Two Subcutaneous Formulations: Vial and Autoinjector (AI) With Olezarsen, at Two Dose Levels, in Healthy Adult Participants
Brief Title: A Study Comparing Two Subcutaneous Formulations: Vial and Autoinjector (AI) With Olezarsen, at Two Dose Levels, in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ISIS 678354-CS20
Expanded Access: NCT06360237 (Approved for marketing)
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Healthy Participants
MeSH Terms: interventions — olezarsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olezarsen Dose Level 1 (Experimental): Participants will receive two doses of Dose Level 1 each, using one of the following two sequences: (i) AI on Day 1 of Treatment Period 1, followed by vial on Day 1 of Treatment Period 2; or (ii) vial on Day 1 of Treatment Period 1, followed by AI on Day 1 of Treatment Period 2. A washout period of 28-42 days will be maintained between the 2 treatment periods.
  Interventions: Drug: Olezarsen
- Olezarsen Dose Level 2 (Experimental): Participants will receive two doses of Dose Level 2 each, using one of the following two sequences: (i) AI on Day 1 of Treatment Period 1, followed by vial on Day 1 of Treatment Period 2; or (ii) vial on Day 1 of Treatment Period 1, followed by AI on Day 1 of Treatment Period 2 A washout period of at least 28 days will be maintained between the 2 treatment periods.
  Interventions: Drug: Olezarsen

INTERVENTIONS:
Drug: Olezarsen — Olezarsen will be administered by SC injection.
  Other Names: ISIS 678354

SUMMARY:
The purpose of the study is to assess the bioequivalence of olezarsen between 2 subcutaneous (SC) formulations [(autoinjector (AI) and vial] at 2 dose levels in healthy adult participants.

DETAILED DESCRIPTION:
This is a Phase 1, single-dose, randomized, open-label, two-period, crossover study in approximately 100 healthy participants. The study will consist of an up to 28-day Screening Period, two treatment periods of 15 days each - with the second treatment period starting 28-42 days after the first begins - and a Post-Treatment Follow-Up Period lasting 91 days after the second treatment period begins. Eligible participants will be randomized to two dose groups (50 mg or 80 mg olezarsen). Participants will be dosed once at the beginning of each treatment period, one time using a single-use AI and one time using a single-use vial. Within each dose group, approximately half of the participants will be dosed with the AI first, with the other participants being dosed with the vial first.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated) and any authorizations required by local law, be able to comply with all study requirements prior to receiving any study drug, and be able to communicate effectively with clinic staff
2. Must be a healthy, adult male or female, 18 to 64 years of age (inclusive), and non-smoking (for at least 6 months prior to first study drug administration)
3. Females must be of non-childbearing potential

Exclusion Criteria:

1. Have a known history or presence of any clinically significant hepatic (e.g., hepatic impairment), renal/genitourinary (e.g., renal impairment), gastrointestinal, cardiovascular, cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological, or hematological disease or condition unless determined as not clinically significant by the PI/sub-investigator

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of olezarsen from time 0 to 336 hours (AUC0-336h) | Up to Day 8 of each of Treatment Periods 1 and 2
Maximum plasma concentration of olezarsen (Cmax) | Up to Day 91 of Treatment Period 2

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No